CLINICAL TRIAL: NCT05309850
Title: Primary Disease Prevention With the Lifestyle Tool
Brief Title: Primary Prevention With the Lifestyle Tool
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Lifestyle2
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Diseases; Type 2 Diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Participants get access to the tool or get assigned to a control group without access
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usage of tool (Experimental): Participants get access to the tool and use it regularly
  Interventions: Behavioral: Lifestyle tool
- Controls on usual care (No Intervention): Participants who get randomized to control cannot access the tool. Development of cardiovascular disease or type 2 diabetes is followed via clinical registries.

INTERVENTIONS:
Behavioral: Lifestyle tool — Regular use of the digital Lifestyle tool
  Arms: Usage of tool

SUMMARY:
In this study participants will be randomized to use a digital lifestyle tool over three years or to a control group without access to the tool. The investigators will prospectively via clinical registries follow the incidence and development of type 2 diabetes and cardiovascular disease in those using the tool regularly and those in the control group.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) and type 2 diabetes (T2D) remain leading cause of death in most European countries, and new strategies for prevention are urgently needed.

Considerable evidence suggest that lifestyle changes can prevent or delay the onset of type 2 diabetes and cardiovascular disease. Modifiable lifestyle factors have been established as key drivers of disease onset and progression.

Many prevention programmes are, however, time-limited and fail to provide continuous support. They also require substantial costs and healthcare resources. Furthermore, accessibility to primary and secondary cardiac prevention programmes is highly variable, as is long-term adherence to lifestyle advice.

In light of this, international associations have emphasized the need for innovative, scalable and cost-effective lifestyle interventions that could be integrated into pre-existing healthcare structures. Digital tools have large potential for clinical utility, but there are several important knowledge gaps. First, data on long-term efficacy is scarce. Second, most studies to date have included only small number of individuals, and there is a need for large randomized controlled studies. Third, cost-effectiveness remains to be demonstrated.

The objective or this study is to evaluate a new web-based tool, developed at the University Gothenburg, Sweden, that aims to support patient autonomy and motivation to make sustainable lifestyle changes.

The investigators will test the hypothesis that individuals who have access to the tool get lower incidence of major cardiovascular events (MACE) and type 2 diabetes or in case they already have diabetes develop improved glucose control compared with control individuals.

The study is an investigator-initiated single-center study conducted over three years.

The tool is web-based and used via a computer or mobile phone. It is used at each individual's preferred pace but participants are recommended to login at least every other week. Every round the participants choose a themes (out of appr. 80 possible covering e.g. food, exercise, stress, self-reflection aspects), which takes appr. 15-30 minutes to complete. Participants then reflect on the content and how it could be implemented in daily life. When returning for next round participants are asked to reflect on any changes done since last time. There is no interaction between individual participants.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* Age above 35 years

Exclusion Criteria:

* type 1 diabetes, MODY or secondary diabetes
* conditions or treatments that in the judgement of the Investigator could affect the study evaluation
* connection with the study team, funders, authorities, universities or other public or private bodies in such a way that specific interests in the study outcomes could be suspected.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90000 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiovascular event | 3 years
  Incidence of major adverse cardiovascular event, defined as cardiovascular death, myocardial infarction, stroke, or hospitalization for heart failure compared between participants regularly using the tool and on usual care.
Incidence of type 2 diabetes | 3 yars
  Incidence of type 2 diabetes defined as random plasma glucose >11.1 mmol/L or fasting glucose >7.0 mmol/L or HbA1C ≥6.5% compared between participants regularly using the tool and on usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Rosengren, Principal Investigator — Göteborg University
Locations (1):
- Skane University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results will be shared after deidentification.
Time Frame: Data will be available after publication.
Access Criteria: To researchers who provide a methodologically sound proposal in order to achieve the aims of that proposal. Proposals should be directed by email to internetverktyg@gu.se